CLINICAL TRIAL: NCT01560416
Title: Randomized Phase II Study of Fulvestrant With or Without Ganetespib in Patients With Hormone Receptor-Positive, Metastatic Breast Cancer
Brief Title: Fulvestrant With or Without Ganetespib in HR+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-477
Record Dates: First submitted 2012-02-21; First posted 2012-03-22 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Metastatic; HR positive; ER positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant; STA 9090

STUDY DESIGN:
Intervention Model Description: Participants were randomized 2:1 B Fulvestrant+Ganetespib:A Fulvestrant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A - Fulvestrant (Active Comparator): Fulvestrant: 500 mg administered by intramuscular injection on days 1 and 15 of cycle 1, day 1 of cycle 2 and each subsequent cycle; cycle duration is 28 days Eligible participants on Arm A were allowed to crossover to Arm B upon disease progression. Treatment continued for Arm A participants until 2nd disease progression.
  Interventions: Drug: Fulvestrant
- Arm B - Fulvestrant+Ganetespib (Active Comparator): Fulvestrant: 500 mg administered by intramuscular injection on days 1 and 15 of cycle 1, day 1 of cycle 2 and each subsequent cycle; cycle duration is 28 days Ganetespib: 200 mg/m2 administered intravenously on days 1, 8 and 15 of each 28 day cycle
  Arm B participants whose disease was at a minimum stable could elect to discontinue ganetespib after 6 cycles or stay on combination treatment until disease progression. Otherwise, Arm B participants taken off ganetespib for toxicity were to remain on single agent fulvestrant until disease progression.
  Interventions: Drug: Fulvestrant; Drug: Ganetespib

INTERVENTIONS:
Drug: Fulvestrant
  Other Names: Faslodex
Drug: Ganetespib
  Other Names: STA9090
  Arms: Arm B - Fulvestrant+Ganetespib

SUMMARY:
Ganetespib is a drug that may stop cancer cells from growing. This drug has been used in other research studies and laboratory experiments. It has also been studied in phase I trials, where the appropriate dosing has been determined. Ganetespib is considered an "HSP90 inhibitor". By blocking HSP90, ganetespib is thought to reduce the ability of cancer cells to become resistant to treatment.

Fulvestrant is a hormonal therapy that works by attaching to estrogen receptors. In doing so, it can block the effect of estrogen on cancer cells. In addition, fulvestrant causes a decrease in the number of estrogen receptors. Fulvestrant is a drug that is approved by the FDA for treatment of metastatic, hormone receptor positive breast cancer, based upon the results of phase III clinical trials.

In the laboratory, adding ganetespib to fulvestrant appears to improve its effectiveness. It is not known whether this is true in humans. In this research study, we are evaluating the effect of the addition of ganetespib to fulvestrant in participants with hormone receptor-positive, metastatic breast cancer.

DETAILED DESCRIPTION:
Because no one knows which of the study options is best, you will be "randomized" into one of the study groups: Arm A: Fulvestrant or Arm B: Fulvestrant plus Ganetespib. You will have a one-third chance of being placed in Arm A and a two-thirds chance of being placed in Arm B.

If you are initially placed in Arm A but your disease progresses, you will have the option of receiving the combination of fulvestrant plus ganetespib as part of Arm C.

You will undergo the following procedures during the research study: study drug(s), blood tests, clinical exams and scans/imaging tests.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer that is metastatic or unresectable locally advanced
* Estrogen and/or progesterone receptor positive breast cancer
* HER2 negative
* Measurable disease is required (effective 4/30/14: all non-measurable [evaluable] disease slots have been filled)
* Endocrine resistant breast cancer
* May have received up to one prior line of chemotherapy for metastatic or unresectable locally advanced breast cancer
* May have initiated bisphosphonate therapy prior to start of protocol therapy
* Must be at least 2 weeks from prior chemotherapy or radiotherapy
* ECOG performance status of 0 or 1
* Availability of tissue block from initial breast cancer diagnosis and/or metastatic recurrence
* For subjects with biopsy-accessible disease, must be willing to undergo a required on-treatment research biopsy
* Adequate IV access

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior treatment with HSP90 inhibitor
* Prior treatment with fulvestrant
* Concurrent treatment with commercial agents or other agents with the intent to treat the participant's malignancy
* Untreated or progressive brain metastases
* Pending visceral crisis, in the opinion of the treating investigator
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fulvestrant or ganetespib
* Uncontrolled intercurrent illness
* Other malignancies within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy U Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - DFCI at Faulkner Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New Hampshire Oncology and Hematology, P.A., Concord, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between June 2012 and June 2015
Period: Randomized Phase
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Started | 15 | 35
Completed | 8 | 35
Not Completed | 7 | 0
Not completed — Crossover Participants | 7 | 0
Period: Crossover Phase
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Started (Only participants randomized to Arm A potentially received crossover treatment.) | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib | Total
Number analyzed (Participants) | 15 | 35 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 29 | 43
  >=65 years | 1 | 6 | 7
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 68] | 52 [31 to 74] | 53 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 34 | 49
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 34 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 30 | 45
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 35 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS based on Kaplan-Meier is defined as the time from study entry to the earliest documentation of disease progression (PD) or death. Participants alive without evidence of PD are censored at the date of last disease assessment. Participants who receive non-protocol anti-cancer therapy before disease progression are censored at time of last disease assessment.
Time Frame: Disease was assessed radiographically every 2 cycles for year 1 and every 2-4 cycles longer-term. Participants in this study cohort were followed for survival up to 4 years from treatment end.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Number analyzed (Participants) | 15 | 35
months | 3.7 [1.0 to 12.0] | 3.6 [2.0 to 7.5]
Statistical Analysis 1: Comparison: ARM A - Fulvestrant vs Arm B - Fulvestrant+Ganetespib; Test type: Superiority; p = 0.79, Log Rank

2. Secondary Outcome: Grade 3-4 Toxicity Rate
Description: All grade 3-4 adverse events (AE) with treatment attribution of possibly, probably or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) as reported on case report forms were counted to calculate the percentage of participants experiencing at least one treatment-related grade 3 or 4 AE of any type on treatment.
Time Frame: AEs were assessed every cycle on treatment (weeks 2-3 on cycle 1). Median treatment duration was 4 cycles/~4 months on each arm. Maximum treatment duration was 41 cycles (Arm A) and 42 cycles (Arm B) which approximates 38 months.
Measure: Number; unit: percentage of participants
Groups:
- Arm A - Crossover Fulvestrant+Ganetespib: Fulvestrant: 500 mg administered by intramuscular injection on days 1 and 15 of cycle 1, day 1 of cycle 2 and each subsequent cycle; cycle duration is 28 days Ganetespib: 200 mg/m2 administered intravenously on days 1, 8 and 15 of each 28 day cycle
  Eligible participants on Arm A were allowed to crossover to Arm B upon disease progression. Treatment continued for Arm A participants until 2nd disease progression.
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib | Arm A - Crossover Fulvestrant+Ganetespib
Number analyzed (Participants) | 15 | 35 | 7
percentage of participants | 100 | 100 | 100

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with measurable disease at baseline achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was assessed radiographically every 2 cycles for year 1 and every 2-4 cycles thereafter on treatment. Maximum treatment duration was 41 cycles (Arm A) and 42 cycles (Arm B) which approximates 38 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Number analyzed (Participants) | 15 | 35
percentage of participants | 20.0 [4.3 to 48.1] | 14.3 [4.8 to 30.3]
Statistical Analysis 1: Comparison: ARM A - Fulvestrant vs Arm B - Fulvestrant+Ganetespib; Test type: Superiority; p = 0.68, Fisher Exact

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with measurable disease at baseline achieving complete response (CR), partial response (PR), or stable disease (SD) for 24 weeks or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria. SD needed to be a minimum 24 weeks in duration.
Time Frame: as for outcome 3
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Number analyzed (Participants) | 15 | 35
percentage of participants | 33.3 [11.8 to 61.6] | 34.3 [19.1 to 52.2]

5. Secondary Outcome: Overall Survival (OS)
Description: OS based on Kaplan-Meier is defined as the time from study entry to death or date last known alive or censored at date last known alive.
Time Frame: Participants were followed long-term for survival every 3 months from the end of treatment until death, lost to follow-up or up to 4 years from treatment end. Median survival follow-up was 28 months for the study cohort.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib
Number analyzed (Participants) | 15 | 35
months | 25.9 [23.1 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI. | 29.2 [26.9 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI.

ADVERSE EVENTS:
Time Frame: AEs were assessed every cycle on treatment (weeks 2-3 on cycle 1). Median treatment duration was 4 cycles/~4 months on each arm. Maximum treatment duration was 41 cycles (Arm A) and 42 cycles (Arm B) which approximates 38 months.
Arm/Group | ARM A - Fulvestrant | Arm B - Fulvestrant+Ganetespib | Arm A - Crossover Fulvestrant+Ganetespib
All-Cause Mortality (participants affected / at risk) | 11/15 | 15/35 | 6/7
Serious Adverse Events (participants affected / at risk) | 2/15 | 11/35 | 0/7
Other Adverse Events (participants affected / at risk) | 15/15 | 35/35 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A - Fulvestrant (N=15) | Arm B - Fulvestrant+Ganetespib (N=35) | Arm A - Crossover Fulvestrant+Ganetespib (N=7)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (7) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Left hand tremors
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Liver bleed
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0)
Infections and infestations-other (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) — Port infection
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A - Fulvestrant (N=15) | Arm B - Fulvestrant+Ganetespib (N=35) | Arm A - Crossover Fulvestrant+Ganetespib (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 34 (34) | 6 (6)
fatigue (General disorders) | 9 (9) | 23 (23) | 2 (2)
nausea (Gastrointestinal disorders) | 6 (6) | 22 (22) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (11) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 10 (10) | 0 (0)
insomnia (Psychiatric disorders) | 2 (2) | 9 (9) | 2 (2)
constipation (Gastrointestinal disorders) | 7 (7) | 8 (8) | 0 (0)
hot flashes (Vascular disorders) | 6 (6) | 8 (8) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8) | 0 (0)
pain (General disorders) | 4 (4) | 8 (8) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 6 (6) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 1 (1)
aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (5) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0)
gastrointestinal disorders-other (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 1 (1)
injection site reaction (General disorders) | 4 (4) | 3 (3) | 0 (0)
non-cardiac chest pain (General disorders) | 2 (2) | 3 (3) | 0 (0)
rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
infections and infestations-other (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT01560416/Prot_SAP_000.pdf